CLINICAL TRIAL: NCT05652608
Title: Stronger Together Psoriatic Arthritis Wellness Study
Status: Recruiting | Type: Observational
Sponsor: Global Healthy Living Foundation (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00062932
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Particpants: participating in Immune Strength, a multi-week wellness program
  Interventions: Behavioral: Immune Strength

INTERVENTIONS:
Behavioral: Immune Strength — Multi-week wellness program provided by the Cleveland Clinic

SUMMARY:
Patients diagnosed with psoriatic arthritis (PsA) confront decisions about how to treat their disease, interact with their health care providers, and modify lifestyle choices that may improve treatment outcomes. With sponsorship support from Janssen and in partnership with the Cleveland Clinic, this survey study will seek to understand and examine whether people living with PsA are interested in and motivated to participate in wellness activities. This cross-sectional observational survey study will help researchers and clinicians to better understand what some of the barriers and facilitators experienced by patients are when considering participation in guided online wellness activities.

People that qualify for the study and complete a 10-minute survey will be invited to participate in Immune Strength, an online wellness program developed by the Cleveland Clinic. Immune Strength is a free 10-week program for creating better habits for a more resilient immune system. By following this program, participants will have the opportunity to learn about how to develop strategies and implement behavior changes for healthier immune functioning.

Participants will be recruited by the Global Healthy Living Foundation (GHLF). GHLF is the parent organization of the CreakyJoints® (CJ) arthritis patient community and primary site for the PCORI-funded Arthritis Patient Partnership with Comparative Effectiveness Researchers (AR-PoWER) Patient Powered Research Network (PPRN), known as ArthritisPower®. ArthritisPower is a subset of CreakyJoints members who have expressed interest in participating in research and signed an informed consent form to participate in the PPRN and its associated research. Any individuals recruited from CreakyJoints or Facebook, who are not already members of ArthritisPower will be encouraged to join the ArthritisPower registry research app, but will not be required to do so in order to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be residents of the United States and United States territories
* Participants must be age 19 and above for United States resident or 21 and above for Puerto Rico residents
* Participants must have a self-reported diagnosis of psoriatic arthritis (PsA) (as indicated by survey screening questions)
* Participants must be taking prescribed medication to treat their PsA
* Participants must have access to a computer or smartphone to take the survey

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by the Global Healthy Living Foundation (GHLF). GHLF is the parent organization of the CreakyJoints® (CJ) arthritis patient community and primary site for PatientSpot Patient Powered Research Network (PPRN), known as PatientSpot®. PatientSpot is a subset of CreakyJoints members who have expressed interest in participating in research and signed an informed consent form to participate in the PPRN and its associated research. Any individuals recruited from CreakyJoints or Facebook, who are not already members of PatientSpot will be encouraged to join the PatientSpot registry research app, but will not be required to do so in order to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Interest in Wellness Programs | Day 1
  Percent of participants interested in participating in a wellness program to complement treatment for controlling their disease
Barriers to Wellness | Day 1
  Percent of participants that experience barriers in using wellness to help manage their disease

CONTACTS AND LOCATIONS:
Locations (1):
- Global Healthy Living Foundation, Upper Nyack, New York, United States

IPD SHARING:
Plan to Share IPD: No